CLINICAL TRIAL: NCT00000374
Title: Preventing Morbidity in First-Episode Schizophrenia
Brief Title: Treatment for First-Episode Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The Zucker Hillside Hospital (Other)
Responsible Party: Principal Investigator, Delbert Robinson, Delbert Robinson, MD/Prinicipal Investigator, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH060004-01 (NIH); R01MH060004-01 (NIH); DSIR 83-ATAP
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Schizophrenia
Keywords: Adolescence; Adult; Antipsychotic Agents; Female; Human; Male; olanzapine; Risperidone; Schizophrenia; Antipsychotic Agents -- *therapeutic use; olanzapine -- *therapeutic use; Risperidone -- *therapeutic use; Schizophrenia -- *drug therapy
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Risperidone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Olanzapine — The dosage for Olanzapine will be 2.5 mg to 20mg per day. The dose of the Olanzapine will be based on the participant's clinical improvement and side effects.
Drug: Risperidone — The dosage for Risperidone will be 1 mg to 6mg per day. The dose of the Risperidone will be based on the participant's clinical improvement and side effects.

SUMMARY:
This 3-year study will determine if the antipsychotic medications olanzapine (Zyprexa®) and risperidone (Risperdal®) can help patients with first-episode schizophrenia.

DETAILED DESCRIPTION:
The goal of the study is to prevent morbidity in first-episode schizophrenia using second-generation antipsychotic drugs: olanzapine, risperidone.

Long-term studies of first-episode schizophrenia patients have clearly indicated excellent initial responsiveness of positive psychotic symptoms to treatment with conventional antipsychotic medications. However, in the years immediately following this initial good response, morbidity increases. Relapses, often multiple ones, are the rule and are usually precipitated by medication noncompliance. There is some evidence that the second-generation antipsychotic drugs may have superior efficacy in terms of these outcome domains. However, these newer agents have been studied primarily in chronic and/or treatment-resistant patient samples and there are virtually no long-term studies or studies comparing the new drugs with one another.

First episode patients are randomly assigned to treatment with olanzapine or risperidone for 3 years. Outcome measures for the initial episode include psychopathology (positive, negative, and affective symptoms), side effects, neurocognition (executive function, memory, and attention), social and occupational function and service utilization. The effects on long-term course are measured in terms of frequency and timing of relapses, level of recovery from subsequent episodes and prospectively assessed course of psychopathology, neurocognitive function, social/vocational function, and service utilization.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00320671

ELIGIBILITY:
Inclusion Criteria:

* First episode schizophrenia, schizophreniform disorder or schizoaffective disorder

Exclusion Criteria:

* Prior treatment with antipsychotic medications.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 1998-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Treatment response | 8 consecutive weeks

CONTACTS AND LOCATIONS:
Overall Officials: Delbert Robinson, MD, Principal Investigator — The Zucker Hillside Hospital
Locations (2):
- United States (2):
  - Hillside Hospital, Glen Oaks, New York
  - Bronx-Lebanon Hospital Center, The Bronx, New York

REFERENCES:
- [Derived] Gallego JA, Robinson DG, Sevy SM, Napolitano B, McCormack J, Lesser ML, Kane JM. Time to treatment response in first-episode schizophrenia: should acute treatment trials last several months? J Clin Psychiatry. 2011 Dec;72(12):1691-6. doi: 10.4088/JCP.10m06349. Epub 2011 Sep 6. PMID 21939612